CLINICAL TRIAL: NCT00896194
Title: Self-Efficacy in Weight Loss Treatment
Acronym: SELF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lora Burke (Other)
Responsible Party: Sponsor-Investigator, Lora Burke, Professor of Nursing and Epidemiology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P01NR010949-PRO08050004; P01NR010949 (NIH)
Record Dates: First submitted 2009-05-07; First posted 2009-05-11 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity; Self-Efficacy; Treatment Adherence
MeSH Terms: conditions — Overweight; Obesity; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Standard Behavioral Treatment (SBT) (Active Comparator): This group receives standard behavioral treatment for weight loss as described below.
  Interventions: Behavioral: Standard Behavioral Treatment
- 2: Modified SBT + Self-Efficacy (Experimental): This group receives modified SBT with an additional self-efficacy component as described below.
  Interventions: Behavioral: Modified Standard Behavioral Intervention + Self-Efficacy

INTERVENTIONS:
Behavioral: Standard Behavioral Treatment — SBT consists of group counseling sessions where participants learn about healthy eating and physical activity. Participants are also given standard calorie goals, fat gram goals, and physical activity goals (minutes).
  Arms: 1: Standard Behavioral Treatment (SBT)
Behavioral: Modified Standard Behavioral Intervention + Self-Efficacy — This group receives identical group intervention sessions. The goals (calories, fat grams, and physical activity minutes) are tailored to the individual's progress. Participants meet regularly with an interventionist for one-on-one lifestyle counseling.
  Arms: 2: Modified SBT + Self-Efficacy

SUMMARY:
This randomized clinical trial of weight loss treatment will examine if adding personalized, one-on-one treatment session to standard behavioral group treatment will result in greater weight loss, less weight regain after weight loss, and better adherence to the treatment protocol.

Everyone who enrolls in the study will receive information on healthy eating, how to increase their physical activity and develop healthy exercise habits and ways to change their eating so that they will lose weight. This information will be provided at evening group sessions. There will be a total of 20 group meetings over an 18-month period that will be held:

* every week during the first month of the study,
* every other week for the second month
* once a month for months 3-12
* every 6 weeks for months 13-18

Participants in the self-efficacy group will also be asked to participate in one-on-one lifestyle counseling sessions with a study interventionist throughout the study.

Everyone will be asked to complete questionnaires, two 24-hour dietary recalls over the phone, and have blood tests done every six months (at the beginning of the study, at 6, 12, and 18 months) a total of 4 times for the study.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* BMI > 27 and < 43
* willing to be randomized to one of the two treatment conditions
* successful completion of screening requiring 5-day recording of food intake in a paper diary
* have at least two risk factors for coronary heart disease, e.g., overweight or obese, hypertension, dyslipidemia, positive family history (first degree relative)

NOTE: Although residing in Western Pennsylvania is not an explicit eligibility criterion, participants are asked to travel to the University of Pittsburgh frequently (weekly for the first month)

Exclusion Criteria:

* presence of a current serious illness or unstable condition requiring physician-supervised diet and exercise (e.g., diabetes, recent acute myocardial infarction) for which physician supervision of diet and physical activity prescription is needed
* physical limitations precluding ability to engage in physical activity at moderate intensity
* pregnancy or intention to become pregnant in the next 18 months
* current treatment for a psychological disorder
* reported alcohol intake > 4 drinks/day
* previous participation in a formal weight loss program within the past 5 years, e.g., Weight Watchers or a research program, or current use of weight loss medication
* planned extended vacations, absences, or relocation within the next 18 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-05; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Weight | 12 and 18 months post enrollment

SECONDARY OUTCOMES:
Health-related quality of life | 12 and 18 months post enrollment
Adherence to treatment protocol | 12 and 18 months post enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Lora E. Burke, PhD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh School of Nursing, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Imes CC, Zheng Y, Mendez DD, Rockette-Wagner BJ, Mattos MK, Goode RW, Sereika SM, Burke LE. Group-Based Trajectory Analysis of Physical Activity Change in a US Weight Loss Intervention. J Phys Act Health. 2018 Nov 1;15(11):840-846. doi: 10.1123/jpah.2017-0484. Epub 2018 Oct 12. PMID 30314417
- [Derived] Zheng Y, Sereika SM, Ewing LJ, Danford CA, Terry MA, Burke LE. Association between Self-Weighing and Percent Weight Change: Mediation Effects of Adherence to Energy Intake and Expenditure Goals. J Acad Nutr Diet. 2016 Apr;116(4):660-6. doi: 10.1016/j.jand.2015.10.014. Epub 2015 Dec 25. PMID 26727241
- [Derived] Goode RW, Ye L, Sereika SM, Zheng Y, Mattos M, Acharya SD, Ewing LJ, Danford C, Hu L, Imes CC, Chasens E, Osier N, Mancino J, Burke LE. Socio-demographic, anthropometric, and psychosocial predictors of attrition across behavioral weight-loss trials. Eat Behav. 2016 Jan;20:27-33. doi: 10.1016/j.eatbeh.2015.11.009. Epub 2015 Nov 14. PMID 26609668